CLINICAL TRIAL: NCT01379495
Title: Randomized Controlled Clinical Trial on Telephone Follow-up in Rehabilitation of Burn Patients: Impact on Health Status
Brief Title: Education Program for Burn Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Natalia Gocalves, RN, PhD student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: uspqueimados2011
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Burns
Keywords: burns; rehabilitation
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Burns victims will receive information according to the service routine
- educational program+telephone follow up (Experimental): Burns victims will participate in an educative program including telephone follow-up during six months after hospital discharge
  Interventions: Behavioral: educational program+telephone follow up

INTERVENTIONS:
Behavioral: educational program+telephone follow up — burns victims will participate in an educative program including telephone follow-up during six months after hospital discharge
  Arms: educational program+telephone follow up

SUMMARY:
The purpose of this study is to assess the effect of an educative program including telephone follow-up for burn patients regarding the impact of this intervention on the health status and return to work at six months after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* adult burned patients (18 years or older), male and female
* patients burned for the first time who needed hospitalization at the Burns Unit
* in cognitive conditions to participate (being able to tell one's address, day of the week and age or birth date)
* in physical conditions to accomplish self-care.

Exclusion Criteria:

* participants burned due to suicide or with previous psychiatric diagnoses or cognitive and psychological difficulties that do not allow them to answer the instrument questions and take care of themselves.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
change from baseline in perceived health status at six months | six months
  The questionnaire "Burns Specific Health Scale- Revised" developed by Blalock; Bunker; De Vellis (1994), adapted by Ferreira et al. (2008) to Brasilian people, will be used to collect the data at six months between groups.

SECONDARY OUTCOMES:
comparison the return to work of burn victims between groups | baseline and six months
  To compare the return to work of burns victims in intervention group with the return to work of burns victims in control group at six months after hospital discharge, proportions will be calculated (returned to work: yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Natália Gonçalves, PhDcandidate, Principal Investigator — University of Sao Paulo; Lidia Ap Rossi, PhD, Study Chair — University of São Paulo at Ribeirão Preto College of Nursing
Locations (1):
- Burns Unit of the University of São Paulo at Ribeirão Preto Hospital das Clínicas, Ribeirão Preto, São Paulo, Brazil